CLINICAL TRIAL: NCT06003426
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled, Phase 3 Study to Evaluate the Efficacy, Safety, and Tolerability of BMS-986278 in Participants With Idiopathic Pulmonary Fibrosis
Brief Title: A Study to Evaluate the Efficacy, Safety, and Tolerability of BMS-986278 in Participants With Idiopathic Pulmonary Fibrosis
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IM027-068
Record Dates: First submitted 2023-08-15; First posted 2023-08-22 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Idiopathic Pulmonary Fibrosis
Keywords: BMS-986278; LPA1 antagonist; IPF; Pulmonary fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis; Pulmonary Fibrosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- BMS-986278 Dose 1 (Experimental)
  Interventions: Drug: BMS-986278
- BMS-986278 Dose 2 (Experimental)
  Interventions: Drug: BMS-986278
- BMS-986278 Placebo (Placebo Comparator)
  Interventions: Drug: BMS-986278 Placebo

INTERVENTIONS:
Drug: BMS-986278 — Specified dose on specified days
  Other Names: Admilparant
  Arms: BMS-986278 Dose 1; BMS-986278 Dose 2
Drug: BMS-986278 Placebo — Specified dose on specified days
  Arms: BMS-986278 Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy, safety, and tolerability of BMS-986278 in participants with Idiopathic Pulmonary Fibrosis.

ELIGIBILITY:
Inclusion Criteria

* Subjects with IPF aged ≥ 40 years at the time of signing the informed consent.
* Diagnosis of IPF within 7 years prior to screening that is supported by centrally read chest high-resolution computed tomography (HRCT) obtained at screening and verification of usual interstitial pneumonia.
* If on pirfenidone or nintedanib, participants must have been on a stable dose for at least 90 days prior to screening.
* If not currently on pirfenidone or nintedanib, participants must not have received either of these medications within 28 days prior to screening.
* Women who are of childbearing potential must have a highly effective form of contraception and must provide a negative urine/serum pregnancy test.
* Men who are sexually active with women of childbearing potential agree to use male barrier contraception.

Exclusion Criteria

* History of stroke or transient ischemic attack within 3 months prior to screening.
* Participants who exhibit symptoms of heart failure at rest.
* Participants who have a current malignancy or a previous malignancy with less than 2 years free of recurrence or a biopsy that is suspicious for malignancy and the possibility of malignancy cannot be reasonably excluded following additional clinical, laboratory, or other diagnostic evaluations.
* Other protocol-defined Inclusion/Exclusion criteria apply.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1255 (Actual)
Dates: Start 2023-09-14 (Actual); Primary Completion 2026-10-26 (Estimated); Study Completion 2026-10-26 (Estimated)

PRIMARY OUTCOMES:
Number of participants that experience spontaneous syncopal events | At approximately 4 weeks
  Cohort 1
Absolute change from baseline in forced vital capacity (FVC) measured in mL | Up to Week 52
  Cohort 2

SECONDARY OUTCOMES:
Number of participants who discontinued treatment due to any low BP-related Adverse Events | Up to approximately 3 years
  Cohort 1
Disease progression | Up to approximately 3 years
  Cohort 2
  Disease progression will be measured by the time to first disease progression event in at least 1 of the following parameters:
  * Absolute percent predicted forced vital capacity (ppFVC) decline of ≥ 10% from baseline
  * Acute exacerbation of pulmonary fibrosis
  * Respiratory-related hospitalization
  * All-cause mortality
Change from baseline in Living with Pulmonary Fibrosis Questionnaire (L-PF) cough domain score | Up to Week 52
  Cohort 2
Change from baseline in L-PF dyspnea domain score | Up to Week 52
  Cohort 2
Change from baseline in walking distance measured in 6-minute walk test (6MWT) | Up to Week 52
  Cohort 2
Time to the first occurrence of any of the components of the composite endpoint: time to first acute exacerbation of pulmonary fibrosis, first Respiratory-related hospitalization, or all-cause mortality | Up to approximately 3 years
  Cohort 2
Time to absolute percent ppFVC decline of ≥ 10% from baseline | Up to approximately 3 years
  Cohort 2
Time to first acute exacerbation of pulmonary fibrosis | Up to approximately 3 years
  Cohort 2
Time to first Respiratory-related hospitalization | Up to approximately 3 years
  Cohort 2
Time to first pulmonary fibrosis-related hospitalization | Up to approximately 3 years
  Cohort 2
Time to death | Up to approximately 3 years
  Cohort 2
Change from baseline in L-PF fatigue domain score | Up to Week 52
  Cohort 2
Change from baseline in L-PF impacts module score | Up to Week 52
  Cohort 2
Change from baseline in cough numeric rating scale (NRS) | Up to Week 52
  Cohort 2
Change from baseline in EuroQol 5 Dimension 5 Level (EQ-5D-5L) health utility index score | Up to Week 52
  Cohort 2
Change from baseline in EQ-5D-5L visual analog scale score | Up to Week 52
  Cohort 2
Rate of decline from baseline in FVC (mL) | Up to Week 52
  Cohort 2
Rate of decline in ppFVC from baseline | Up to Week 52
  Cohort 2
Change in ppFVC from baseline | Up to Week 52
  Cohort 2
Proportion of participants with absolute decline in ppFVC ≥10% | Up to Week 52
  Cohort 2
Proportion of participants with relative decline in ppFVC ≥10% | Up to Week 52
  Cohort 2
Change from baseline in single-breath diffusing capacity of the lung for carbon monoxide (DLCO SB) (corrected for hemoglobin) (mL/min/mm Hg) | Up to Week 52
  Cohort 2
Change in percent predicted single breath diffusing capacity of the lung for carbon monoxide (ppDLCO SB) (corrected for hemoglobin) from baseline | Up to Week 52
  Cohort 2
Change from baseline in quantitative lung fibrosis (QLF) score via high-resolution computed tomography (HRCT) | Up to Week 52
  Cohort 2
Number of participants with Adverse Events (AEs) | Up to 28 days after last dose
  Cohort 2
Number of participants with Serious AEs (SAEs) | Up to 28 days after last dose
  Cohort 2
Number of participants with AEs leading to early discontinuation of investigational medicinal product (IMP) | Up to 28 days after last dose
  Cohort 2
Number of participants with AEs related to IMP | Up to 28 days after last dose
  Cohort 2
Number of treatment-emergent deaths | Up to 28 days after last dose
  Cohort 2
Number of participants with clinical laboratory abnormalities | Up to 28 days after last dose
  Cohort 2
Number of participants with electrocardiogram (ECG) abnormalities | Up to 28 days after last dose
  Cohorts 1 and 2
Number of participants with vital sign abnormalities | Up to 28 days after last dose
  Cohorts 1 and 2
Number of participants with physical examination abnormalities | Up to 28 days after last dose
  Cohort 1

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (390):
- United States (70):
  - Local Institution - 0189, Birmingham, Alabama
  - Local Institution - 0361, Phoenix, Arizona
  - Local Institution - 0396, La Jolla, California
  - Local Institution - 0193, Los Angeles, California
  - Local Institution - 0398, Los Angeles, California
  - Local Institution - 0389, Orange, California
  - Local Institution - 0405, Sacramento, California
  - Local Institution - 0185, San Francisco, California
  - Local Institution - 0186, Stanford, California
  - Local Institution - 0363, Aurora, Colorado
  - Local Institution - 0194, Denver, Colorado
  - Local Institution - 0175, New Haven, Connecticut
  - Local Institution - 0151, Newark, Delaware
  - Local Institution - 0367, Washington D.C., District of Columbia
  - Local Institution - 0101, Brandon, Florida
  - Local Institution - 0436, Clearwater, Florida
  - Local Institution - 0425, DeBary, Florida
  - Local Institution - 0079, Gainesville, Florida
  - Local Institution - 0352, Hialeah, Florida
  - Local Institution - 0370, Kissimmee, Florida
  - Local Institution - 0502, Leesburg, Florida
  - Local Institution - 0153, Loxahatchee Groves, Florida
  - Local Institution - 0187, Ocala, Florida
  - Local Institution - 0418, Pensacola, Florida
  - Local Institution - 0206, St. Petersburg, Florida
  - Local Institution - 0364, Tampa, Florida
  - Local Institution - 0372, Dublin, Georgia
  - Local Institution - 0178, Chicago, Illinois
  - Local Institution - 0183, Chicago, Illinois
  - Local Institution - 0058, Chicago, Illinois
  - Local Institution - 0085, Maywood, Illinois
  - Local Institution - 0325, Peoria, Illinois
  - Local Institution - 0180, Iowa City, Iowa
  - Local Institution - 0204, Kansas City, Kansas
  - Local Institution - 0393, Louisville, Kentucky
  - Local Institution - 0354, Baltimore, Maryland
  - Local Institution - 0380, Boston, Massachusetts
  - Local Institution - 0040, Boston, Massachusetts
  - Local Institution - 0472, Ann Arbor, Michigan
  - Local Institution - 0096, Chesterfield, Missouri
  - Local Institution - 0174, St Louis, Missouri
  - Local Institution - 0154, Mount Kisco, New York
  - Local Institution - 0433, Durham, North Carolina
  - Local Institution - 0366, Wilmington, North Carolina
  - Local Institution - 0368, Winston-Salem, North Carolina
  - Local Institution - 0201, Cincinnati, Ohio
  - Local Institution - 0197, Columbus, Ohio
  - Local Institution - 0417, Toledo, Ohio
  - Local Institution - 0181, Oklahoma City, Oklahoma
  - Local Institution - 0373, Tulsa, Oklahoma
  - Local Institution - 0021, Portland, Oregon
  - Local Institution - 0067, Hershey, Pennsylvania
  - Local Institution - 0406, Philadelphia, Pennsylvania
  - Local Institution - 0388, Philadelphia, Pennsylvania
  - Local Institution - 0199, Philadelphia, Pennsylvania
  - Local Institution - 0202, Pittsburgh, Pennsylvania
  - Local Institution - 0346, Wynnewood, Pennsylvania
  - Local Institution - 0375, Anderson, South Carolina
  - Local Institution - 0188, Charleston, South Carolina
  - Local Institution - 0400, Nashville, Tennessee
  - Local Institution - 0073, Dallas, Texas
  - Local Institution - 0377, Dallas, Texas
  - Local Institution - 0039, Houston, Texas
  - Local Institution - 0097, Houston, Texas
  - Local Institution - 0029, McKinney, Texas
  - Local Institution - 0048, San Antonio, Texas
  - Local Institution - 0027, Salt Lake City, Utah
  - Local Institution - 0184, Richmond, Virginia
  - Local Institution - 0191, Everett, Washington
  - Local Institution - 0362, Seattle, Washington
- Argentina (16):
  - Local Institution - 0131, Mar del Plata, Buenos Aires
  - Local Institution - 0019, Buenos Aires, B
  - Local Institution - 0172, Caba, B
  - Local Institution - 0170, Florida, B
  - Local Institution - 0286, Mar del Plata, B
  - Local Institution - 0485, Quilmes, Provincia de Buenos Aires, B
  - Local Institution - 0290, San Juan Bautista, B
  - Local Institution - 0288, Ciudad Autónoma Buenos Aires, C
  - Local Institution - 0287, Godoy Cruz, M
  - Local Institution - 0013, Mendoza, M
  - Local Institution - 0356, Mendoza, M
  - Local Institution - 0330, Rosario, S
  - Local Institution - 0169, San Miguel de Tucumán, T
  - Local Institution - 0218, Córdoba, X
  - Local Institution - 0283, Buenos Aires
  - Local Institution - 0173, Santa Fe
- Australia (10):
  - Local Institution - 0209, Camperdown, New South Wales
  - Local Institution - 0239, Westmead, New South Wales
  - Local Institution - 0210, Brisbane, Queensland
  - Local Institution - 0229, Greenslopes, Queensland
  - Local Institution - 0421, South Brisbane, Queensland
  - Local Institution - 0309, Adelaide, South Australia
  - Local Institution - 0443, Box Hill, Victoria
  - Local Institution - 0420, Frankston, Victoria
  - Local Institution - 0419, Murdoch, Western Australia
  - Local Institution - 0385, Nedlands, Western Australia
- Austria (4):
  - Local Institution - 0458, Salzburg, Salzburger Land
  - Local Institution - 0409, Linz, Upper Austria
  - Local Institution - 0025, Vienna
  - Local Institution - 0459, Vienna
- Belgium (5):
  - Local Institution - 0332, Yvoir, Namur
  - Local Institution - 0075, Brussels
  - Local Institution - 0345, Kortrijk
  - Local Institution - 0038, Leuven
  - Local Institution - 0046, Liège
- Brazil (12):
  - Local Institution - 0084, Belo Horizonte, Minas Gerais
  - Local Institution - 0098, Belo Horizonte, Minas Gerais
  - Local Institution - 0490, Barra Mansa, Rio de Janeiro
  - Local Institution - 0359, Rio de Janeiro, Rio de Janeiro
  - Local Institution - 0304, Porto Alegre, Rio Grande do Sul
  - Local Institution - 0049, Porto Alegre, Rio Grande do Sul
  - Local Institution - 0307, Porto Alegre, Rio Grande do Sul
  - Local Institution - 0089, Blumenau, Santa Catarina
  - Local Institution - 0054, Santo André, São Paulo
  - Local Institution - 0305, São Bernardo do Campo, São Paulo
  - Local Institution - 0024, São Paulo, São Paulo
  - Local Institution - 0486, São Paulo
- Canada (14):
  - Local Institution - 0062, Sherwood Park, Alberta
  - Local Institution - 0100, Kelowna, British Columbia
  - Local Institution - 0061, Vancouver, British Columbia
  - Local Institution - 0171, Vancouver, British Columbia
  - Local Institution - 0103, Burlington, Ontario
  - Local Institution - 0216, Hamilton, Ontario
  - Local Institution - 0044, Owen Sound, Ontario
  - Local Institution - 0213, Toronto, Ontario
  - Local Institution - 0426, Greenfield Park, Quebec
  - Local Institution - 0434, Montreal, Quebec
  - Local Institution - 0215, Québec, Quebec
  - Local Institution - 0495, Saint-Charles-Borromée, Quebec
  - Local Institution - 0053, Trois-Rivières, Quebec
  - Local Institution - 0478, Trois-Rivières, Quebec
- Chile (6):
  - Local Institution - 0503, Concepción, Bio Bio
  - Local Institution - 0437, Curicó, Maule Region
  - Local Institution - 0211, Talca, Maule Region
  - Local Institution - 0051, Quillota, Región de Valparaíso
  - Local Institution - 0068, Santiago, RM
  - Local Institution - 0214, Santiago, RM
- China (42):
  - Local Institution - 0263, Hefei, AH
  - Local Institution - 0222, Hefei, AH
  - Local Institution - 0410, Hefei, Anhui
  - Local Institution - 0238, Beijing, Beijing Municipality
  - Local Institution - 0470, Beijing, BJ
  - Local Institution - 0257, Beijing, BJ
  - Local Institution - 0242, Guangzhou, GD
  - Local Institution - 0480, Guangzhou, Guangdong
  - Local Institution - 0295, Shenzhen, Guangdong
  - Local Institution - 0492, Shenzhen Shi, Guangdong
  - Local Institution - 0294, Zhengzhou, HA
  - Local Institution - 0360, Zhengzhou, HA
  - Local Institution - 0233, Shijiazhuang, HE
  - Local Institution - 0482, Yichang Shi, HE
  - Local Institution - 0369, Wuhan, Hubei
  - Local Institution - 0252, Wuhan, HUB
  - Local Institution - 0424, Suzhou, Jiangsu
  - Local Institution - 0262, Wuxi, Jiangsu
  - Local Institution - 0483, Xuzhou, JS
  - Local Institution - 0431, Nanchang, JX
  - Local Institution - 0479, Shenyang, Liaoning
  - Local Institution - 0241, Shenyang, LN
  - Local Institution - 0292, Shenyang, LN
  - Local Institution - 0255, Shanghai, SH
  - Local Institution - 0230, Shanghai, SH
  - Local Institution - 0243, Chengdu, Sichuan
  - Local Institution - 0391, Tianjin, Tianjin Municipality
  - Local Institution - 0365, Tianjin, Tianjin Municipality
  - Local Institution - 0488, Hangzhou, Zhejiang
  - Local Institution - 0351, Ningbo, Zhejiang
  - Local Institution - 0249, Hangzhou, ZJ
  - Local Institution - 0244, Changsha
  - Local Institution - 0371, Chengdu
  - Local Institution - 0258, Guangzhou
  - Local Institution - 0237, Hohhot
  - Local Institution - 0403, Jinan
  - Local Institution - 0358, Nanjing
  - Local Institution - 0266, Shanghai
  - Local Institution - 0408, Shanghai
  - Local Institution - 0232, Shanghai
  - Local Institution - 0261, Shijiazhuang
  - Local Institution - 0374, Xi'an
- Colombia (6):
  - Local Institution - 0297, Medellín, ANT
  - Local Institution - 0291, Bogotá, DC
  - Local Institution - 0278, Floridablanca, Santander Department
  - Local Institution - 0268, Santiago de Cali, VAC
  - Local Institution - 0138, Bogotá
  - Local Institution - 0279, Manizales
- Denmark (3):
  - Local Institution - 0064, Aarhus, Central Jutland
  - Local Institution - 0010, Odense C, Region Syddanmark
  - Local Institution - 0036, Hellerup
- Finland (2):
  - Local Institution - 0350, Turku, Laensi-Suomen Laeaeni
  - Local Institution - 0328, Helsinki
- France (12):
  - Local Institution - 0047, Bron, Auvergne-Rhône-Alpes
  - Local Institution - 0322, Grenoble, Auvergne-Rhône-Alpes
  - Local Institution - 0083, Nantes, Pays de la Loire Region
  - Local Institution - 0334, Marseille, Provence-Alpes-Côte d'Azur Region
  - Local Institution - 0012, Angers
  - Local Institution - 0066, Bobigny
  - Local Institution - 0321, Brest
  - Local Institution - 0052, Dijon
  - Local Institution - 0022, Paris
  - Local Institution - 0342, Pessac
  - Local Institution - 0023, Toulouse
  - Local Institution - 0339, Tours
- Germany (15):
  - Local Institution - 0050, Freiburg I. Breisgau, Baden-Wurttemberg
  - Local Institution - 0272, Munich, Bavaria
  - Local Institution - 0042, Münnerstadt, Bavaria
  - Local Institution - 0313, Hamburg, Hamburg
  - Local Institution - 0041, Immenhausen, Hesse
  - Local Institution - 0026, Marburg, Hesse
  - Local Institution - 0092, Essen, North Rhine-Westphalia
  - Local Institution - 0320, Cologne, Northwest
  - Local Institution - 0349, Berlin, State of Berlin
  - Local Institution - 0003, Berlin, State of Berlin
  - Local Institution - 0037, Ahrensburg
  - Local Institution - 0004, Coswig
  - Local Institution - 0383, Heidelberg
  - Local Institution - 0017, Leipzig
  - Local Institution - 0347, Mainz
- Greece (6):
  - Local Institution - 0314, Marousi, Attica
  - Local Institution - 0318, Pylaia-Chortiatis, B
  - Local Institution - 0110, Athens
  - Local Institution - 0108, Corfu
  - Local Institution - 0102, Larissa
  - Local Institution - 0109, Rio
- Hungary (2):
  - Local Institution - 0018, Budapest
  - Local Institution - 0343, Győr
- India (18):
  - Local Institution - 0430, Ahmedabad, Gujarat
  - Local Institution - 0282, Surat, Gujarat
  - Local Institution - 0264, Belagavi, Karnataka
  - Local Institution - 0386, Bhopal, Madhya Pradesh
  - Local Institution - 0395, Nagpur, Maharashtra
  - Local Institution - 0414, Nagpur, Maharashtra
  - Local Institution - 0275, Pune, Maharashtra
  - Local Institution - 0498, Pune, Maharashtra
  - Local Institution - 0457, Pune, Maharashtra
  - Local Institution - 0285, New Delhi, National Capital Territory of Delhi
  - Local Institution - 0429, New Delhi, National Capital Territory of Delhi
  - Local Institution - 0428, Mohali, Punjab
  - Local Institution - 0289, Jaipur, Rajasthan
  - Local Institution - 0477, Lucknow, Uttar Pradesh
  - Local Institution - 0247, Dehradun, Uttarakhand
  - Local Institution - 0225, Kolkata, West Bengal
  - Local Institution - 0256, Bangalore
  - Local Institution - 0228, Lucknow
- Ireland (3):
  - Local Institution - 0168, Drogheda, LH
  - Local Institution - 0497, Dublin
  - Local Institution - 0117, Dublin
- Israel (6):
  - Local Institution - 0331, Haifa, HA
  - Local Institution - 0348, Haifa
  - Local Institution - 0113, Jerusalem
  - Local Institution - 0319, Petah Tikva
  - Local Institution - 0035, Rehovot
  - Local Institution - 0090, Tel Aviv
- Italy (17):
  - Local Institution - 0329, Bologna, BO
  - Local Institution - 0326, Modena, Emilia-Romagna
  - Local Institution - 0034, Florence, FI
  - Local Institution - 0119, Milan, MI
  - Local Institution - 0127, Pisa, PI
  - Local Institution - 0005, Roma, RM
  - Local Institution - 0095, Ancona
  - Local Institution - 0118, Bergamo
  - Local Institution - 0057, Foggia
  - Local Institution - 0126, Forlì
  - Local Institution - 0069, Milan
  - Local Institution - 0121, Monza
  - Local Institution - 0323, Napoli
  - Local Institution - 0125, Palermo
  - Local Institution - 0122, Pavia
  - Local Institution - 0120, Sassari
  - Local Institution - 0114, Siena
- Japan (35):
  - Local Institution - 0107, Chiba, Chiba
  - Local Institution - 0088, Fukuoka, Fukuoka
  - Local Institution - 0442, Fukuoka, Fukuoka
  - Local Institution - 0129, Koriyama-shi, Fukushima
  - Local Institution - 0059, Naka-gun, Gunma
  - Local Institution - 0355, Hiroshima, Hirohima-ken
  - Local Institution - 0132, Sapporo, Hokkaido
  - Local Institution - 0031, Himeji-Shi, Hyōgo
  - Local Institution - 0030, Kobe, Hyōgo
  - Local Institution - 0353, Matsusaka-shi, Mie-ken
  - Local Institution - 0077, Nagasaki, NGS
  - Local Institution - 0106, Ginowan-Shi, Okinawa
  - Local Institution - 0299, Osakasayama-shi, Osaka
  - Local Institution - 0274, Sakai, OSK
  - Local Institution - 0123, Hamamatsu, Shizuoka
  - Local Institution - 0105, Bunkyō City, TKY
  - Local Institution - 0009, Shimotsuge-shi, Tochigi
  - Local Institution - 0124, Bunkyo-Ku, Tokyo
  - Local Institution - 0226, Bunkyo-ku, Tokyo
  - Local Institution - 0302, Mitaka-shi, Tokyo
  - Local Institution - 0251, Shinjuku-Ku, Tokyo
  - Local Institution - 0301, Fukuoka
  - Local Institution - 0111, Iizuka-shi
  - Local Institution - 0130, Izumo-Shi
  - Local Institution - 0011, Kamogawa-Shi
  - Local Institution - 0086, Kumamoto
  - Local Institution - 0033, Minatoku
  - Local Institution - 0300, Minatoku
  - Local Institution - 0045, Nagoya
  - Local Institution - 0015, Seto
  - Local Institution - 0074, Shinjyu-Ku
  - Local Institution - 0056, Tenri-Shi
  - Local Institution - 0128, Tokyo
  - Local Institution - 0298, Yokohama
  - Local Institution - 0260, Yoshida-Gun
- Mexico (3):
  - Local Institution - 0324, Metepec, Edo de Mexico
  - Local Institution - 0382, Morelia, Michoacán
  - Local Institution - 0167, Oaxaca City, Oaxaca
- Netherlands (4):
  - Local Institution - 0394, Rotterdam, South Holland
  - Local Institution - 0379, Amsterdam
  - Local Institution - 0152, Heerlen
  - Local Institution - 0456, Nieuwegein
- Peru (3):
  - Local Institution - 0220, Lima, LIM
  - Local Institution - 0144, San Miguel, LIM
  - Local Institution - 0007, Lima
- Poland (6):
  - Local Institution - 0143, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Local Institution - 0145, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Local Institution - 0147, Bialystok, Podlaskie Voivodeship
  - Local Institution - 0333, Gdansk, Pomeranian Voivodeship
  - Local Institution - 0306, Olsztyn, Warmian-Masurian Voivodeship
  - Local Institution - 0159, Lodz
- Portugal (8):
  - Local Institution - 0002, Faro
  - Local Institution - 0139, Lisbon
  - Local Institution - 0142, Lisbon
  - Local Institution - 0028, Lisbon
  - Local Institution - 0134, Loures
  - Local Institution - 0137, Porto
  - Local Institution - 0165, Porto
  - Local Institution - 0158, Vila Nova de Gaia
- Local Institution - 0198, Guaynabo, PR, Puerto Rico
- South Korea (16):
  - Local Institution - 0240, Goyang-si, Gyeonggi-do
  - Local Institution - 0271, Goyang-si, Gyeonggi-do
  - Local Institution - 0224, Jongno-gu, Seoul
  - Local Institution - 0276, Yongsan-gu, Seoul
  - Local Institution - 0441, Dong-gu, Ulsan
  - Local Institution - 0404, Bucheon-si
  - Local Institution - 0227, Bucheonsi Weonmigu
  - Local Institution - 0440, Busan
  - Local Institution - 0284, Donggu
  - Local Institution - 0250, Gyeonggi-do
  - Local Institution - 0231, Haeundae-Gu
  - Local Institution - 0246, Iksansi
  - Local Institution - 0269, Incheon
  - Local Institution - 0265, Seoul
  - Local Institution - 0221, Seoul
  - Local Institution - 0273, Suwon, Gyeonggi-do
- Spain (14):
  - Local Institution - 0093, Santander, CB
  - Local Institution - 0140, Santiago de Compostela, C
  - Local Institution - 0099, Madrid, M
  - Local Institution - 0065, Madrid, M
  - Local Institution - 0161, Madrid, M
  - Local Institution - 0149, Majadahonda, M
  - Local Institution - 0135, Barcelona
  - Local Institution - 0341, Barcelona
  - Local Institution - 0166, Girona
  - Local Institution - 0496, Madrid
  - Local Institution - 0338, Madrid
  - Local Institution - 0155, Madrid
  - Local Institution - 0146, Oviedo
  - Local Institution - 0335, Pamplona
- Switzerland (3):
  - Local Institution - 0160, Basel, Canton of Basel-City
  - Local Institution - 0461, Bern, Canton of Bern
  - Local Institution - 0473, Geneva, Canton of Geneva
- Taiwan (9):
  - Local Institution - 0491, Changhua, CHA
  - Local Institution - 0481, Kaohsiung City, Kao-Hsiung
  - Local Institution - 0484, Taichung, TXG
  - Local Institution - 0235, Douliu Shi, YUN
  - Local Institution - 0259, Kaohsiung City
  - Local Institution - 0270, New Taipei City
  - Local Institution - 0267, Taichung
  - Local Institution - 0254, Taipei
  - Local Institution - 0236, Taipei
- Turkey (Türkiye) (8):
  - Local Institution - 0176, Gümüşhane, Gümüşhane Province
  - Local Institution - 0177, Ankara
  - Local Institution - 0150, Bursa
  - Local Institution - 0205, Izmir
  - Local Institution - 0207, Izmir
  - Local Institution - 0196, Maltepe
  - Local Institution - 0200, Pasaport
  - Local Institution - 0344, Topkapı
- United Kingdom (11):
  - Local Institution - 0378, Birmingham, BIR
  - Local Institution - 0415, Bristol, BST
  - Local Institution - 0402, Cambridge, Cambridgeshire
  - Local Institution - 0164, Dundee, DND
  - Local Institution - 0072, Edinburgh, EDH
  - Local Institution - 0337, London, Greater London
  - Local Institution - 0407, Oxford, Oxfordshire
  - Local Institution - 0336, Peterborough, PTE
  - Local Institution - 0416, Cottingham, Yorkshire and the Humber
  - Local Institution - 0411, Birmingham
  - Local Institution - 0438, Leeds

IPD SHARING:
Plan to Share IPD: Yes
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria. Additional information regarding Bristol Myer Squibb's data sharing policy and process can be found at: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See plan description
Access Criteria: See plan description
URL: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsclinicaltrials.com/us/en/clinical-trials/NCT06003426.html